CLINICAL TRIAL: NCT04740944
Title: The Effect of Salutogenic Approach Based Interview on Sense of Coherence and Psychological Resistance of People With Schizophrenia: A Randomized Controlled Trial
Brief Title: Salutogenic Approach Based Interview With People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Özgür Sema ACI, Dr, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Nurse_Psychiatric
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Salutogenesis; Mental Health Disorder; Schizophrenia; Sense of Coherence
Keywords: Salutogenesis; sense of coherence; resilience; schizophrenia
MeSH Terms: conditions — Mental Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): the intervention group was subjected to salutogenic approach-based interview consisting of 16 sessions twice a week.
  Interventions: Behavioral: Salutogenic Approach Based Interview
- Control group (No Intervention): The control group continued their routine activities and was interviewed face-to-face 5 times.

INTERVENTIONS:
Behavioral: Salutogenic Approach Based Interview — Salutogenic Approach Based Interview has five basic components. (1) Continuity of health, (2) The story of the person, (3) Health promoting factors, (4) Understanding the health promoting power of tension and strain, (5) Active adaptation In traditional therapy recommended for recovery, more emphasis is placed on negative life events, diagnosis and medication. In the salutogenic approach-based interview, the resources and coping potential of the person are discussed and three healing factors are focused on for the recovery process. These factors are that the participants (1) perceive themselves as more than just a diagnosis and disease, (2) self-discovery and respect for other people's self-discovery, (3) control over their own lives. In the intervention, mental health nurses take part as group leaders. The focus in interviews is therapeutic conversations.
  Arms: Intervention group

SUMMARY:
This study determines the effectiveness of the interviewing based on salutogenic approach on the sense of coherence and resilience of people with schizophrenia. For this, while the intervention group was subjected to salutogenic approach-based interview consisting of 16 sessions twice a week. The control group continued their routine activities and was interviewed face-to-face 5 times.

DETAILED DESCRIPTION:
Schizophrenia is a chronic and serious disease that affecting 20 million people in the world. Because of the problems these individuals face in cognitive, emotional, and behavioral domains, they have frequently difficulty in adapting to their environment, have to struggle against stigmatization, have an increased risk of committing suicide due to ever decreasing functioning and hopelessness they experience, and they need a long-term care and support due to their difficulty in compliance to treatment.

The sense of coherence and resilience are important components for individuals diagnosed with schizophrenia to cope with problems in cognitive, emotional, and behavioral domains. Sense of coherence reflects the capacity of a person to respond stressful situations. It is associated with a person's emotional responses and resources, making sense of the world, use of required resources, and respond to demands. Powerful sense of coherence helps a person to protect own health, to cope with the stress factors, to manage the strain, and to activate their resources.

Resilience is described as the capacity of individuals to recover or adapt after problems, difficult periods, and stressful life crises that they face during their life. This term can also be understood as the ability to ensure and/or maintain a state of coherence.

The model addressing the concepts of sense of coherence and resilience is salutogenic model. Salutogenic model (1996) which was developed by Aaron Antonovsky (1923-1994) is an alternative model to pathogenesis approach. While pathogenesis focuses on how the disease has occurred, salutogenesis focuses on how wellbeing is formed. Salutogenic approach attempts to explain why some people better cope with the strain, stressful life events and difficulties they face and how they maintain their health and wellbeing better compared to others. The most significant factor in personal evaluation of an external stimulus and in coping with the strain is explained with sense of coherence which is specified in the model. Sense of coherence is the fundamental concept of salutogenic theory and consists of three components. These are comprehensibility, manageability, and meaningfulness. Comprehensibility expresses that internal and external stressors experienced by a person are "expected" and "explainable" in the life. Manageability is the sense about that individual has the internal and external resources to cope with the situation caused by stressor. Meaningfulness states a person's perception on how they struggle against negative life events.

Lindström and Eriksson (2010) describe salutogenesis as an "umbrella". Under this umbrella, there are also concepts of "empowerment", "self-efficacy", "quality of life", "resilience", "welfare", and "competence" as well as the sense of coherence. It is accepted that all of these concepts are associated with salutogenic dimensions and provide significant contributions to describe, explain, analyze, and promote health.

There are studies applying intervention programs based on salutogenic model in people with mental disorder or groups at risk in terms of mental disorder. The first intervention program based on salutogenic model is talk therapy. The major goal of this application is to increase awareness and confidence of the participants and to promote their sense of coherence, coping skills, mental health, and welfare level by allowing them to recognize internal/external resources and potentials. With the talk therapy application, it is provided to manage stressful situations effectively by bringing out personal and collective resistance resources.

The intervention based on salutogenic model has five fundamental components. (1) Sustainability of health, (2) Story of the person, (3) Factors to promote health, (4) Understanding the health promotion power of tension and strain, (5) Active adaptation.

Traditional therapy which is recommended for recovery focuses on negative life events, diagnosis, and medication. In the talk therapy based on salutogenic approach, resources and coping potential of a person are addressed and three recovery factors are focused for the recovery process. These factors are (1) participants' perception about themselves as more than only a diagnosis and disease, (2) getting respected about discovering themselves and getting discovered by other people, (3) having control of their own lives. Psychiatric nurses take part as group leaders in the intervention. Focus of the talk therapies is their speech.

It is stated that it could be possible for a person diagnosed with schizophrenia to gradually regain the ability of functioning independently, to rebuild family relationships, and to fulfil professional roles and functions with the practices to be made by the help of salutogenic model. Therefore, these people should be empowered to decide about their lives. By this means, it is possible to lead a satisfying life for them against the restrictions caused by the disease. A study evaluating sense of coherence and quality of life for people diagnosed with schizophrenia revealed that sense of coherence was an indicator for the quality of life. Bengtsson-Tops and Hansson (2001) concluded in their literature review on sense of coherence that the studies using methods regarding care, support and recovery of people diagnosed with schizophrenia or schizoaffective disorder could be useful in terms of recovery. In the light of these findings, Bengtsson-Tops and Hansson concluded that actions to improve cognitive abilities of people in order to facilitate the recovery could be increased by the concepts of sense of coherence. Menzies (2000) providing detailed information about how salutogenic approach should be applied for a person diagnosed with schizophrenia highlighted that psychiatric nurse would develop a person's hopes allowing them to cope with symptoms and problems, would enhance their self-esteem supporting their abilities and skills, would contribute development of their personal identity, and would increase the sense of coherence.

It is stated in the literature that practices based on salutogenic model and talk therapy based on this model could be used for people diagnosed with schizophrenia. In the international literature, there is no study in which salutogenic-based talk therapy program is applied to only people diagnosed with schizophrenia. In Turkey, there has been no study examining the efficacy of any intervention program based on this model.

ELIGIBILITY:
Inclusion criteria of the study:

* Getting diagnosed with schizophrenia or schizoaffective disorder
* Completing acute treatment and being at maintenance medication period

Exclusion criteria of the study

* Being at the period of psychotic relapse
* Having mental development disorder
* Being under the influence of alcohol-drugs
* Having diagnosed with personal disorder
* Being considered unsuitable to include in the group study by doctors and nurses of CMHC.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Sense of Coherence Scale_13 (SOC_13) | 8 weeks
  At the end of 8 weeks (16 sessions of salutogenic approach based interview ), they were evaluated using the sense of coherence scale which was developed by Antonovsky (1987) is a self-report scale consisting of a total of 13 items ranging between 1 and 7. The scale allows to use subscale scores and calculate total score. Higher scale scores indicate that individual has higher sense of coherence. In the reliability studies of the original version of the scale, internal consistency coefficients were calculated as .62 for "meaningfulness", .54 for "manageability", .57 for "comprehensibility", and .69 for overall scale.
Brief Resilience Scale (BRS) | 8 weeks
  At the end of 8 weeks (16 sessions of salutogenic approach based interview ), they were evaluated using brief resilience scale which was developed by Smith et al., (2008) to measure resilience of individuals. The scale is a 5-point likert self-report assessment instrument with 6 items. High BRS scores signify higher resilience of a person.

SECONDARY OUTCOMES:
Sense of Coherence Scale_13 (SOC_13) | 12 weeks
  At the end of 12 weeks (16 sessions of salutogenic approach based interview + 1 month), they were evaluated using the sense of coherence scale which was developed by Antonovsky (1987) is a self-report scale consisting of a total of 13 items ranging between 1 and 7. The scale allows to use subscale scores and calculate total score. Higher scale scores indicate that individual has higher sense of coherence. In the reliability studies of the original version of the scale, internal consistency coefficients were calculated as .62 for "meaningfulness", .54 for "manageability", .57 for "comprehensibility", and .69 for overall scale.
Brief Resilience Scale (BRS) | 12 weeks
  At the end of 8 weeks (16 sessions of salutogenic approach based interview ), they were evaluated using brief resilience scale which was developed by Smith et al., (2008) to measure resilience of individuals. The scale is a 5-point likert self-report assessment instrument with 6 items. High BRS scores signify higher resilience of a person.

CONTACTS AND LOCATIONS:
Overall Officials: OZGUR S ACI, Dr, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa Institute of Granduate Studies, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share to IPD

REFERENCES:
- [Background] Arvidsdotter T, Marklund B, Taft C, Kylen S. Quality of life, sense of coherence and experiences with three different treatments in patients with psychological distress in primary care: a mixed-methods study. BMC Complement Altern Med. 2015 Apr 26;15:132. doi: 10.1186/s12906-015-0654-z. PMID 25928131
- [Background] Badura-Brzoza K, Zajac P, Matysiakiewicz J, Piegza M, Rycerski W, Hese RT, Koczy B, Semenowicz J. [The association of quality of life with mental status and sociodemographic data in patients after total hip replacement]. Psychiatr Pol. 2008 Mar-Apr;42(2):261-9. Polish. PMID 19697531
- [Background] Bag B, Salutogenic model in mental health and psychiatric nursing. Current Approaches in Psychiatry. 2017:9: 284-300.
- [Background] Baş AU, Yurdabakan İ. The predictive value of resilience and school climate in life satisfaction among middle school students. Mehmet Akif Ersoy University Journal of Education Faculty. 2017;1: 202-214.
- [Background] Bengtsson-Tops A, Brunt D, Rask M. The structure of Antonovsky's sense of coherence in patients with schizophrenia and its relationship to psychopathology. Scand J Caring Sci. 2005 Sep;19(3):280-7. doi: 10.1111/j.1471-6712.2005.00342.x. PMID 16101857
- [Background] Bengtsson-Tops A, Hansson L. The validity of Antonovsky's Sense of Coherence measure in a sample of schizophrenic patients living in the community. J Adv Nurs. 2001 Feb;33(4):432-8. doi: 10.1046/j.1365-2648.2001.01692.x. PMID 11251730
- [Background] Bilge A, Mermer G, Çam O, Çetinkaya A, Erdoğan E, Üçkuyu N. Profıle of communıty mental health centers in Turkey between 2013-2015 years. Journal of Health Sciences of Kocaeli University. 2016;(2): 1-5.
- [Background] Çapan BE, Arıcıoğlu A. Forgiveness as predictor of psychological resiliency. e-International Journal of Educational Research. 2014;(5): 70-82.
- [Background] Doğan T. Adaptation of the brief resilience scale into Turkish: A validity and reliability study. The Journal of Happiness ve Well-Being. 2015;3: 93-102.
- [Background] Eriksson M. The Sense of Coherence in the Salutogenic Model of Health. 2016 Sep 3. In: Mittelmark MB, Sagy S, Eriksson M, Bauer GF, Pelikan JM, Lindstrom B, Espnes GA, editors. The Handbook of Salutogenesis [Internet]. Cham (CH): Springer; 2017. Chapter 11. Available from http://www.ncbi.nlm.nih.gov/books/NBK435812/ PMID 28590620
- [Background] Gassmann W, Christ O, Lampert J, Berger H. The influence of Antonovsky's sense of coherence (SOC) and psychoeducational family intervention (PEFI) on schizophrenic outpatients' perceived quality of life: a longitudinal field study. BMC Psychiatry. 2013 Jan 7;13:10. doi: 10.1186/1471-244X-13-10. PMID 23294596
- [Background] Griffiths CA. Sense of coherence and mental health rehabilitation. Clin Rehabil. 2009 Jan;23(1):72-8. doi: 10.1177/0269215508095360. PMID 19114439
- [Background] Griffiths CA. A critical analysis of Antonovsky's sense of coherence theory in relation to mental health and mental disorder and the effect of a lifelong learning intervention on the sense of coherence of mental health service users, Doktoral Thesis, Middlesex University.Dubai. 2010.
- [Background] Hjelle EG, Bragstad LK, Kirkevold M, Zucknick M, Bronken BA, Martinsen R, Kvigne KJ, Kitzmuller G, Mangset M, Thommessen B, Sveen U. Effect of a dialogue-based intervention on psychosocial well-being 6 months after stroke in Norway: A randomized controlled trial. J Rehabil Med. 2019 Sep 3;51(8):557-565. doi: 10.2340/16501977-2585. PMID 31411337
- [Background] Izydorczyk B, Sitnik-Warchulska K, Kuhn-Dymecka A, Lizinczyk S. Resilience, Sense of Coherence, and Coping with Stress as Predictors of Psychological Well-Being in the Course of Schizophrenia. The Study Design. Int J Environ Res Public Health. 2019 Apr 9;16(7):1266. doi: 10.3390/ijerph16071266. PMID 30970589
- [Background] Jakovljevic M. Empathy, Sense of Coherence and Resilience: Bridging Personal, Public and Global Mental Health and Conceptual Synthesis. Psychiatr Danub. 2018 Dec;30(4):380-384. doi: 10.24869/psyd.2018.380. PMID 30439796
- [Background] Jensen BB, Dur W, Buijs G. The Application of Salutogenesis in Schools. 2016 Sep 3. In: Mittelmark MB, Sagy S, Eriksson M, Bauer GF, Pelikan JM, Lindstrom B, Espnes GA, editors. The Handbook of Salutogenesis [Internet]. Cham (CH): Springer; 2017. Chapter 22. Available from http://www.ncbi.nlm.nih.gov/books/NBK435853/ PMID 28590654
- [Background] Kasperek-Zimowska B, Chadzynska M. [Sense of coherence and coping styles among parents of adult children with schizophrenia]. Psychiatr Pol. 2011 Sep-Oct;45(5):643-52. Polish. PMID 22220482
- [Background] Korlin D, Wrangsjo B. Treatment effects of GIM therapy. Nordic Journal of Music Therapy. 2002.(11): 3-15.
- [Background] Köroğlu A, Hocaoğlu Ç. The effect of schizophrenia on the family. Journal of Duzce Univertsity Health Sciences Institute. 2017;(7): 170-175.
- [Background] Langeland E, Sense of coherence and life satisfaction in people suffering from mental health problems. An intervention study in talk-therapy groups with focus on salutogenesis. Doctoral Thesis, Dissertation for The Degree Doctor Rerum Politicarum, University of Bergen, Norway.(2007).
- [Background] Langeland E, Riise T, Hanestad BR, Nortvedt MW, Kristoffersen K, Wahl AK. The effect of salutogenic treatment principles on coping with mental health problems A randomised controlled trial. Patient Educ Couns. 2006 Aug;62(2):212-9. doi: 10.1016/j.pec.2005.07.004. Epub 2005 Oct 19. PMID 16242903
- [Background] Langeland E, Vinje HF. The Application of Salutogenesis in Mental Healthcare Settings. 2016 Sep 3. In: Mittelmark MB, Sagy S, Eriksson M, Bauer GF, Pelikan JM, Lindstrom B, Espnes GA, editors. The Handbook of Salutogenesis [Internet]. Cham (CH): Springer; 2017. Chapter 28. Available from http://www.ncbi.nlm.nih.gov/books/NBK435815/ PMID 28590623
- [Background] Menzies V. Depression in schizophrenia: nursing care as a generalized resistance resource. Issues Ment Health Nurs. 2000 Sep;21(6):605-17. doi: 10.1080/01612840050110308. PMID 11271136
- [Background] Petavy F, Guizzaro L, Antunes Dos Reis I, Teerenstra S, Roes KCB. Beyond "Intent-to-treat" and "Per protocol": Improving assessment of treatment effects in clinical trials through the specification of an estimand. Br J Clin Pharmacol. 2020 Jul;86(7):1235-1239. doi: 10.1111/bcp.14195. Epub 2020 Mar 27. PMID 31883123
- [Background] Schrank B, Brownell T, Jakaite Z, Larkin C, Pesola F, Riches S, Tylee A, Slade M. Evaluation of a positive psychotherapy group intervention for people with psychosis: pilot randomised controlled trial. Epidemiol Psychiatr Sci. 2016 Jun;25(3):235-46. doi: 10.1017/S2045796015000141. Epub 2015 Feb 20. PMID 25698298
- [Background] Tan KK, Chan SWC, Vehviläinen-Julkunen K. Self-care program for older Community-dwellers: protocol for a randomized controlled trial. Central European Journal of Nursing and Midwifery. 2014; 5(4): 145-155.
- [Background] Veltro F, Nicchiniello I, Pica A, Pontarelli I, Iannone C, Pontarelli C, Zappone L, Vendittelli N. [Description and impact of a structured psychoeducational and salutogenetic approach (InteGRO) to support the recovery of people with severe mental disorders]. Riv Psichiatr. 2018 Jul-Aug;53(4):205-213. doi: 10.1708/2954.29697. Italian. PMID 30087491
- [Background] Witkowska-Luc B. Schizophrenia and sense of coherence. Psychiatr Pol. 2018 Apr 30;52(2):217-226. doi: 10.12740/PP/OnlineFirst/69697. Epub 2017 Jun 29. English, Polish. PMID 29975362
- [Result] Forsberg KA, Bjorkman T, Sandman PO, Sandlund M. Influence of a lifestyle intervention among persons with a psychiatric disability: a cluster randomised controlled trail on symptoms, quality of life and sense of coherence. J Clin Nurs. 2010 Jun;19(11-12):1519-28. doi: 10.1111/j.1365-2702.2009.03010.x. Epub 2010 Apr 5. PMID 20384660
- See also: WHO (2019) World Health Report — https://www.who.int/news-room/fact-sheets/detail/mental-disorders